CLINICAL TRIAL: NCT02802969
Title: Improvement of Local Control in Skull Base, Spine and Sacral Chordomas Treated by Surgery and Protontherapy Targeting Hypoxic Cells Revealed by [18F]FAZA) PET/CT Tracers
Acronym: PROTONCHORDE01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IC 2014-16
Record Dates: First submitted 2016-06-03; First posted 2016-06-16 (Estimated); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Skull Base Chordoma; Vertebral Chordoma
MeSH Terms: interventions — Surgical Procedures, Operative; fluoroazomycin arabinoside

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- [18F]FAZA PET/CT (Experimental): In residual chordoma tumors after surgery, Investigators propose a protontherapy guided by conventional imaging (CT/MRI) and a boost guided by FAZA PET/CT, in order to target the hypoxic zones and to increase the dose in an adequate manner, which could result in improving long-term local control and reducing complications.
  Interventions: Procedure: Surgery; Radiation: Protontherapy; Drug: 18F FAZA

INTERVENTIONS:
Procedure: Surgery — The operative approach and operating time will be performed according to neurosurgical practices (for head and neck) or surgical orthopaedic team (for sacrum) depending on the location, the extension and the relationship of the lesion to critical structures.
  The surgery can be macroscopically complete or incomplete.
Radiation: Protontherapy — Radiotherapy will be done with the Cyclotron, for a total dose of 78 Gray Relative Biological Effective (Gy RBE) - 70 Gy RBE to the tumor bed and macroscopic volume and 8 Gy RBE to the the hypoxic component volume, delivered in 39 fractions spread over 67 days.
Drug: 18F FAZA — FAZA PET/CT, in order to target the hypoxic zones
  Other Names: 18F FLUOROAZOMYCIN-ARABINOFURANOSIDE

SUMMARY:
Improved local control of chordoma initially treated with surgery or not, thanks to adjuvant radiotherapy oriented by conventional imaging Computed Tomography /Magnetic Resonance Imaging (CT / MRI) and guided by the [18Fluor] ([18F]) Fluoroazomycin Arabinofuranoside (FAZA) Positron Emission Tomography / Computed Tomography (PET / CT) to target the radioresistant hypoxic cells.

DETAILED DESCRIPTION:
Due to the close contacts of the lesion with the neurovascular structures, in the case of skull base chordoma and mobile spine, surgery is often incomplete. On the contrary, surgery of the sacral region (for which the block excision is often possible) brings a better therapeutic outcome. Radiotherapy with high-dose supplement improves the outcomes for all these lesions.

Intratumoral hypoxia is a primary factor of radioresistance, it's known since long by radiation oncologists. [18F]FAZA gives an image of the hypoxic volume target. Investigators propose to increase the radioactive dose in the hypoxic volume target but in order to succeed, radiation oncologists have to precisely identify this hypoxic volume. Radiation oncologists would increase of 10% the radioactive dose that will allow us to improve local control at 3 years of 15% without any additional side effect.

ELIGIBILITY:
Inclusion Criteria:

* Typical chordoma and chondroid chordoma of the skull base, spine or chordoma of sacral region
* Patient undergoing an additional or exclusive radiotherapy (Photontherapy and/or Prothontherapy)
* Age ≥ 18 years old
* ECOG performance status 0 to 2
* Satisfying biological functions 28 days before inclusion :

  1. Haemoglobin ≥ 9 g/dL
  2. Neutrophils ≥ 1500/mm3
  3. Platelets ≥ 100 000/mm3
  4. ASAT, ALAT, GGT, PAL ≤ 1.5 N, bilirubin ≤ 40 μmol/L, LDH ≤ 1.5 N
  5. Creatininemia < 1.5 N
* Satisfying vital cardiac and respiratory functions
* Neurologic functions well stabilised
* Effective contraception for women of childbearing age during the the protontherapy treatment and during the month following the end of treatment. A pregnancy test shall be negative at inclusion.
* Patient covered by health insurance
* Patient provided with information and signature of informed consent.

Exclusion Criteria:

* Dedifferentiated chordomas, chondrosarcoma
* History of cancer (except cutaneous basocellular epithelioma or epithelioma of the uterine cervix) having recurred in the 5 years preceding entry in the trial and no relapse in the last 3 years
* Metastatic patient
* History of brain radiation therapy, or base of the skull or spinal segments to be treated
* Contraindications to radiotherapy
* Contraindications to PET/CT examinations [18F] Fluorodexoxyglucose (FDG) and [18]FAZA
* Associated pathology likely to prevent the patient from receiving treatment,
* Incompatible treatment with the inclusion in the study (oxygen therapy, EPO, anti-vascular treatments, anti-angiogenic treatments)
* Patient already included in another therapeutic trial with an experimental medication,
* Patient currently nursing,
* Persons deprived of their liberty, or under guardianship,
* Impossibility of undergoing the trial's medical follow-up for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-07-22 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
Improvement local control of chordomas according to RECIST criteria. | 36 months
  Rate of local control at 3 years
Improvement local control of chordomas according to PERCIST criteria | 36 months
  Rate of local control at 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Hamid MAMMAR, MD, Principal Investigator — Institut Curie
Locations (1):
- Institut Curie - Hôpital René Huguenin, Saint-Cloud, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share de-identified data sets with interested researchers, educators or clinicians. Materials generated under the project will be disseminated in accordance with Institut Curie policies.
Time Frame: Data requests can be submitted starting 9 months after article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific reserach, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).